CLINICAL TRIAL: NCT07243132
Title: Long-Terms Responders in Metastatic Lung Cancer: Better Understanding for Better Management (LUNGEVITY STUDY)
Acronym: LUNGEVITY
Status: Recruiting | Type: Observational
Sponsor: GFPC Investigation (Other)
Responsible Party: Sponsor
Organization: Groupe Francais De Pneumo-Cancerologie (Other)
Other Study IDs: GFPC INVESTIGATION 07-2019
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-08

CONDITIONS: Metastatic Lung Cancer; Metastatic NSCLC; Metastatic Small Cell Lung Cancer
Keywords: long-terms responders; Mestastatic Lung Cancer; Metastatic NSCLC; Metastatic small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma | interventions — 4-amino-4'-hydroxylaminodiphenylsulfone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Long-Terms Responders in metastatic Lung Cancer: Long-term responders defined as patients alive for three years after diagnosis of metastatic Lung cancer (NSCLC and SCLC) and not receiving cytotoxic chemotherapy at the time of inclusion.
  Interventions: Behavioral: Hospital Anxiety and Depression scale (HAD); Behavioral: Quality of Life Questionnaire - Lung Cancer 13 (QLQ-LC13); Behavioral: Questionnaire Aix-Marseille-Université (AMU)

INTERVENTIONS:
Behavioral: Hospital Anxiety and Depression scale (HAD) — The HAD scale is an instrument used to screen for anxiety and depressive disorders. It comprises 14 items rated from 0 to 3. Seven questions relate to anxiety (total A) and seven others to depression (total D), giving two scores (maximum score for each = 21).
Behavioral: Quality of Life Questionnaire - Lung Cancer 13 (QLQ-LC13) — The EORTC QLQ-LC13: a 13-item lung cancer-specific questionnaire module supplement to the EORTC core quality of life questionnaire (QLQ-C30) for use in lung cancer clinical trials. The QLQ-LC13 includes questions assessing lung cancer-associated symptoms (cough, haemoptysis, dyspnoea and site specific pain), treatment-related side effects (sore mouth, dysphagia, peripheral neuropathy and alopecia) and pain medication.
Behavioral: Questionnaire Aix-Marseille-Université (AMU) — Data analysis will be firstly descriptive in order to report on the quality of life of respondents. Then, in a second stage, the factors associated with quality of life will be analyzed using linear or logistic regression models depending on the nature of the variable of interest.

SUMMARY:
The goal of this observational study is to identify and describe the clinical characteristics, health status, socio-economic impacts and quality of life of patients alive for three years after diagnosis of metastatic Lung cancer and no longer receiving cytotoxic chemotherapy. The main question is to identify the needs of these patients in terms of health status (impact of cancer treatments, incidence of new diseases, cardiovascular, diabetes, second cancers), socio-economic aspects, quality of life and return to employment.

Participants will be asked to answer quality of life questionnaires at the time of inclusion and 6 and 12 months after inclusion and then, every year up to 5 years in this study.

They will be followed regularly, in consultations, according to the usual practices of the physicians in each participating center.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old
* Patients alive after more than three years from diagnosis with stage IV or Stage III NSCLC or SCLC, not treated with cytotoxic chemotherapy at the time of inclusion (the patient may be undergoing imunotherapy, targeted therapy or surveillance).
* Patients covered by the French National Health Insurance program or with thirdparty-payer health insurance

Exclusion Criteria:

* Difficulties for understanding French
* Patients undergoing treatment with cytotoxic chemotherapy
* Patients under legal guardianship, under curatorship or tutorship
* Insufficient cognitive capacity to answer questions
* Inability to obtain data collection (lost to follow-up, patient's refusal for data collection)
* Patients refusing the collection of their data (an information sheet will be provided)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited by GFPC centers which is a large French network of hospitals and clinics particularly active in pneumology and thoracic oncology centers participating in clinical research.
  The principal investigator in each center will identify consecutive patients eligible for inclusion. Patients will be asked to confirm their consent for data collection.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-07-02 (Actual); Primary Completion 2031-01-31 (Estimated); Study Completion 2031-01-31 (Estimated)

PRIMARY OUTCOMES:
Baseline Clinical Characteristics | At Baseline visit, on a maximum period of 12 months.
  Metastatic Lung Cancer Long-Terms Responders clinical characteristics: baseline patient demographics, clinical and pathological characteristics (e.g. age, medical history, comorbidities, past history of cancer, smoking status, NSCLC or SCLC characteristics)
Aix-Marseille-University (AMU) questionnaire | At inclusion, 6 and 12 months after inclusion and every year up to 5 years
EORTC QLQ-LC13 | at inclusion, 6 and 12 months after inclusion and every year up to 5 years
Hospital Anxiety and Depression Scale (HAD) | at inclusion, 6 and 12 months after inclusion and every year up to 5 years
Treatment characteristics | From date of first lung cancer treatment administration up to 5 years
  Treatment characteristics are defined by the type of treatment, the numbers of cycle and the duration of treatment.
Health status | At Baseline visit and up to 5 years
  Health status will be evaluated using Eastern Cooperative Oncology Group performance status (PS), and collecting data new diseases, cardiovascular, diabetes, second cancers
Socio-demographic characteristics | At Baseline visit and up to 5 years
  Socio-demographic characteristics will be evaluated based on the following data: professional, socio-family and socio-economic characteristics, education, family status, potential professional exposure(s)

SECONDARY OUTCOMES:
Progression free survival (PFS) | From date of first lung cancer treatment administration up to 5 years
  PFS is defined as the length of time during and after the treatment of cancer, that a patient lives with the disease but it does not get worse. PFS will be assessed by local review, as per the current practice at site.
Overall Survival (OS) | From date of first lung cancer treatment initiation up to 5 years
  Overall Survival is defined as the length of time from the start of treatment for the cancer that patients diagnosed with the disease are still alive.

CONTACTS AND LOCATIONS:
Overall Officials: Lionel FALCHERO, Principal Investigator — GFPC; Laurence BIGAY-GAME, Principal Investigator — GFPC
Locations (45):
- France (45):
  - CH du Pays d Aix, Aix-en-Provence
  - CHU Angers, Angers
  - Hôpital Henri Duffaut, Avignon
  - CH Bastia, Bastia
  - APHP Hôpital Avicennes, Bobigny
  - CHU Morvan, Brest
  - Hôpital Louis Pradel, Bron
  - Pneumologie Centre François Baclesse, Caen
  - Centre Hospitalier du Cotentin, Cherbourg
  - CHU Hôpital Montpied, Clermont-Ferrand
  - Oncologie CLCC Jean Perrin, Clermont-Ferrand
  - Pneumologie Hospices Civils de Colmar, Colmar
  - Pneumologie Centre Hospitalier Intercommunal de Créteil, Créteil
  - Centre Hospitalier d'Elbeuf - Pneumologie, Elbeuf
  - CH Eure-Seine, Évreux
  - Grand Hôpital de l'Est Francilien - Site Marne la Vallée, Jossigny
  - Centre Hospitalier Les Oudairies, La Roche-sur-Yon
  - CH La Rochelle, La Rochelle
  - Hôpital Robert Boulin, Libourne
  - Hôpital de la Vallée, Longjumeau
  - Hôpital du Scorff, Lorient
  - Pneumologie Hôpital privé Jean Mermoz, Lyon
  - Centre Léon Bérard, Lyon
  - Hôpital Européen, Marseille
  - Hôpital Nord - Oncologie Thoracique, Marseille
  - GHEF Site de Meaux, Meaux
  - CHRU de Nancy, Nancy
  - CHU Nantes, Nantes
  - Pneumologie Hôpital Cochin, Paris
  - Hôpital Tenon, Paris
  - Hôpital La Pitié-Salpêtrière, Paris
  - Pneumologie Centre Hospitalier, Pau
  - Centre Catalan d'Oncologie, Perpignan
  - CHU Reims Hôpital Maison Blanche, Reims
  - CHU Hôpital Ponchailloux, Rennes
  - Hôpital Charles Nicolle, Rouen
  - Hôpital Privé de la Loire, Saint-Etienne
  - Pneumologie CHU St Etienne, Saint-Etienne
  - CH des Vallées de l'Ariège, Saint-Jean-de-Verges
  - CHU La Réunion Site Sud, Saint-Pierre
  - CH de Saint Malo, St-Malo
  - Hôpital d'Instruction des Armées Saint-Anne, Toulon
  - Hôpital Larrey, Toulouse
  - Oncologie CH Bretagne-Atlantique, Vannes
  - Centre Hospitalier de Villefranche sur Saone, Villefranche-sur-Saône

IPD SHARING:
Plan to Share IPD: Undecided